CLINICAL TRIAL: NCT03756740
Title: The Effectiveness of Telerehabilitation Modalities in Physical Therapy in the Management of Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Principal Investigator, Gali Dar, principal investigator, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 196/18
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Low Back Pain
Keywords: telerehabilitation, exercises, video, physical therapy
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Telerehabilitation; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Sixty patients diagnosed with chronic LBP referred for physical therapy to one of the 5 outpatient clinics of Maccabi Health Services in the Haifa metropolitan area, Israel, will be recruited for this study. each subject will undergo a baseline examination including answering several questionnaires/self-reported outcome measures, a history of present or any past LBP and a physical examination routinely conducted during physical therapy assessment and treatments.
  Following the physical examination, the physical therapist will decide on the appropriate physical therapy modalities for the specific patients. These techniques will include only manual therapy (soft tissue mobilization and vertebrae segmental mobilization) and interferential electrotherapy. Furthermore, the subject will receive an appropriate exercise program which will performed at home.
  Each subject will be randomly referred to one of the research groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know the intervention in other groups or the research aim in details. they will only know that it is a research for low back pain treatment.
  The physical therapists performing the examination pre and post intervention will be blinded to the participants group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): After each face to face session the patient will receive the exercises ordered by the physical therapist to perform at home. The exercises will be sent as a video to his/her mobile or e-mail according to the subject's preference. The exercises will be previously recorded and accompanied with a verbal explanation and instructions on how to correctly perform the exercises, paying close attention to specific points. In total, there will be 10 videos of exercises found effective for LBP patients.. After each face to face meeting, the physical therapist will choose from these 10 videos suitable exercises for the patients.
  Interventions: Other: telerehabilitation and physical therapy
- Control (Active Comparator): After each face to face session the patient will receive the exercises ordered by the physical therapist to perform at home.
  subjects will receive the same exercises given to experimental group according to the results of the face to face meeting. The exercises will be shown as printed pictures on paper
  Interventions: Other: control

INTERVENTIONS:
Other: telerehabilitation and physical therapy — subject will receive the LBP exercises as a video to his/her mobile or e-mail
  Arms: Telerehabilitation
Other: control — subjects will receive the LBP exercises as printed pictures on paper
  Arms: Control

SUMMARY:
Low back pain (LBP), a common disorder, causes disability, functional decline and high health care costs. Patient care programs include specific exercises for promoting function and improving health. Self-practice and adherence to treatment are important for treatment success and better outcomes. Telerehabilitation (TR) might improve patient symptoms, compliance to treatment and reduce patient symptoms, however, its effectiveness in treating LBP, still needs further investigation.

The overall aim of this study will be to examine the effectiveness of combining telerehabilitation within physical therapy treatments for patients with LBP

DETAILED DESCRIPTION:
The study will include 60 patients complaining of chronic nonspecific LBP over a 6 month period of time and referred for physical therapy treatment. They will undergo a routine physical examination and be assigned a personal treatment (manual therapy and electrotherapy) and exercise program in accordance with their condition. Participants will receive a total of 8 treatments over a 4-week period (twice a week).

The sample will be randomly divided into 2 groups: a. research group A will receive a video of the exercises via e-mails or to their cellphones; b. a control group will receive the exercises printed on paper.

The exercises will be recorded and be supplemented by a verbal explanation and instructions as to how to correctly perform the exercises. In total, there will be ten videos, found to be important and effective for LBP patients. From these videos, a physical therapist will choose the most suitable exercises for the patients after each treatment meeting (face to face). The patients will be assessed at baseline, at the end of treatment and at a 3 month follow-up telephone assessment.

ELIGIBILITY:
Inclusion Criteria:

* Main complaint of nonspecific LBP over a 3 month period
* Possess a smartphone, e-mail and the understanding of using these tools for viewing videos.

Exclusion Criteria:

* Signs or symptoms of possible malignancy are present, such as unexplained weight loss, slight or no reduction of pain while in a recumbent position or subjects were not screened prior to referral to physical therapy.
* two or more of the following signs are present on physical examination: lower extremity weakness in a myotome distribution, decreased sensation in a dermatomal distribution, altered lower extremity deep tendon reflexes, pathological reflexes, a positive straight leg raise (SLR) test, crossed SLR or femoral nerve stretch test.
* Symptoms began immediately after a significant trauma (motor vehicle accident, fall from a height) and subjects were not been screened for possible fractures.
* Physical therapy or chiropractic treatment for LBP was provided during the 6 months prior to participation in the study or are currently being treated.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 3 months
  level of pain on an 11-point numeric pain rating scale
Modified Oswestry Disability Index | 3 months
  questionnaire to assess the disability level associated with LBP and includes 10 questions regarding activities likely to be affected by LBP
Fear-Avoidance Beliefs Questionnaire | 3 months
  questionnaire to assess the subject's beliefs as to the potential harm of several physical and work-related activities
Survey Health Form Short | 3 months
  questionnaire to assess the subject's belief as to his/her health-related quality of life

SECONDARY OUTCOMES:
Global rating of change | 3 months
  a 15-point Likert scale ranging to assess treatment success
A questionnaire regarding treatment satisfaction | 3 months
  a 5-point Likert scale to assess patient satisfaction from treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, PhD, Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
following study completion, a paper will be submitted to international professional journal
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months following end of study